CLINICAL TRIAL: NCT00443534
Title: A Treatment Protocol For Patients Continuing From A Prior SU011248 Protocol.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6181078
Record Dates: First submitted 2007-03-02; First posted 2007-03-06 (Estimated); Results first posted 2013-05-24 (Estimated); Last update posted 2013-05-24 (Estimated); Status verified 2013-04

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: SU011248

INTERVENTIONS:
Drug: SU011248 — Administered orally in doses ranging from 25 to 50 mg once daily; dosing schedule and dosage depends on the patients dosing from the prior protocol
  Other Names: Sutent/Sunitinib

SUMMARY:
This protocol allows subjects who have participated in a previous SU011248 protocol the ability to continue to receive SU011248 after their study has ended.

ELIGIBILITY:
Inclusion Criteria:

* Participation in a previous SU011248 protocol and are judged by the investigator to have the potential to derive clinical benefit by remaining on SU011248 after the prior protocol ends.

Exclusion Criteria:

* Severe acute or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2006-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (54):
- United States (32):
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Littleton, Colorado
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Harvey, Illinois
  - Pfizer Investigational Site, Maywood, Illinois
  - Pfizer Investigational Site, Tinley Park, Illinois
  - Pfizer Investigational Site, Zion, Illinois
  - Pfizer Investigational Site, Munster, Indiana
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Grand Rapids, Michigan
  - Pfizer Investigational Site, City of Saint Peters, Missouri
  - Pfizer Investigational Site, Creve Coeur, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Hackensack, New Jersey
  - Pfizer Investigational Site, Chapel Hill, North Carolina
  - Pfizer Investigational Site, Clinton, North Carolina
  - Pfizer Investigational Site, Goldsboro, North Carolina
  - Pfizer Investigational Site, Hickory, North Carolina
  - Pfizer Investigational Site, Wilson, North Carolina
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Hershey, Pennsylvania
  - Pfizer Investigational Site, Greenville, South Carolina
  - Pfizer Investigational Site, Greer, South Carolina
  - Pfizer Investigational Site, Spartanburg, South Carolina
  - Pfizer Investigational Site, Bedford, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Fort Worth, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, San Antonio, Texas
- Canada (3):
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Ottawa, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
- France (3):
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Villejuif
- Germany (4):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Großhansdorf
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Wiesbaden
- Italy (6):
  - Pfizer Investigational Site, Bologna
  - Pfizer Investigational Site, Cremona
  - Pfizer Investigational Site, Genova
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Orbassano (TO)
  - Pfizer Investigational Site, Rozzano (MI)
- Spain (3):
  - Pfizer Investigational Site, Elche, Alicante
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Córdoba, Cordoba
- United Kingdom (3):
  - Pfizer Investigational Site, Sutton, Surrey
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Manchester

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181078&StudyName=A%20Treatment%20Protocol%20For%20Patients%20Continuing%20From%20A%20Prior%20SU011248%20Protocol.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited from following previous sunitinib trials: NCT00798889, NCT00092001, NCT00137449, A6181049, A6181051, NCT00113516, NCT00265317, NCT00137423, NCT00267748, NCT00243503, NCT00471276, NCT00174434, NCT00528619, NCT00372775, NCT00417885, NCT00428597, and NCT00372567.
Groups:
- Sunitinib: Participants received sunitinib (SU011248) capsules in one of the standard sunitinib schedules: Schedule 4/2 [4 weeks on study drug, 2 weeks off treatment]; Schedule 2/1 [2 weeks on study drug, 1 week off treatment]; Schedule 2/2 [2 weeks on study drug, 2 weeks off treatment]; or continuous dosing). The starting dose for all dosing regimens except continuous dosing was 50 milligram (mg) orally once daily (37.5 mg orally once daily for continuous dosing).
Period: Overall Study
Arm/Group | Sunitinib
Started | 123
Treated | 122
Completed | 0
Not Completed | 123
Not completed — Lack of Efficacy | 67
Not completed — Adverse Event | 16
Not completed — Death | 9
Not completed — Withdrawal by Subject | 8
Not completed — Study Terminated by Sponsor | 12
Not completed — Other | 10
Not completed — Enrolled, Not Treated | 1

BASELINE CHARACTERISTICS:
Arm/Group | Sunitinib
Number analyzed (Participants) | 122
Age Continuous [Mean (Standard Deviation); unit: years] | 59.9 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 61

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Baseline up to Day 28 after last dose of study treatment
Population: Intent to treat (ITT) population included all enrolled participants who received at least 1 dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 122
participants
  Adverse Events | 119
  Serious Adverse Events | 35

2. Other Pre Specified Outcome: Overall Survival (OS)
Description: Time in weeks from the start of study treatment to date of death due to any cause. OS was calculated as (the death date minus the date of first dose of study medication plus 1) divided by 7. Death was determined from adverse event data (where outcome was death) or from follow-up contact data (where the participant current status was death).
Time Frame: Baseline, every 2 months until death or up to 2 years after the last dose of study treatment
Population: Tumor response data were not formally analyzed in this study as individual participant outcomes contributed to conclusions in their prior studies.
Arm/Group | Sunitinib
Number analyzed (Participants) | 0

3. Other Pre Specified Outcome: Progression-Free Survival (PFS)
Description: Time in weeks from start of study treatment to first documentation of objective tumor progression or death due to any cause. PFS was calculated as (first event date minus the date of first dose of study medication plus 1) divided by 7. Tumor progression was determined from oncologic assessment data (where data meet the criteria for progressive disease [PD]), or from adverse event (AE) data (where the outcome was "Death").
Time Frame: Baseline, every 2 months until objective tumor progression or death or up to 2 years after the last dose of study medication
Population: as for outcome 2
Arm/Group | Sunitinib
Number analyzed (Participants) | 0

4. Other Pre Specified Outcome: Time to Tumor Progression (TTP)
Description: Time in weeks from start of study treatment to first documentation of objective tumor progression or death due to cancer, whichever comes first. TTP was calculated as (first event date minus the date of first dose of study medication plus 1) divided by 7. Tumor progression was determined from oncologic assessment data (where data meet the criteria for progressive disease [PD]).
Time Frame: Baseline, every 2 months until objective tumor progression or up to 2 years after the last dose of study medication
Population: as for outcome 2
Arm/Group | Sunitinib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Sunitinib
Serious Adverse Events (participants affected / at risk) | 35/122
Other Adverse Events (participants affected / at risk) | 115/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=122)
Anaemia (Blood and lymphatic system disorders) | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 1
Congestive cardiomyopathy (Cardiac disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2
Small intestinal obstruction (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Chest pain (General disorders) | 1
Condition aggravated (General disorders) | 1
Disease progression (General disorders) | 9
Gait disturbance (General disorders) | 1
Oedema peripheral (General disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 2
Appendicitis perforated (Infections and infestations) | 1
Biliary sepsis (Infections and infestations) | 1
Catheter site infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 2
Dehydration (Metabolism and nutrition disorders) | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Hypertensive emergency (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=122)
Anaemia (Blood and lymphatic system disorders) | 24
Leukopenia (Blood and lymphatic system disorders) | 7
Neutropenia (Blood and lymphatic system disorders) | 32
Thrombocytopenia (Blood and lymphatic system disorders) | 17
Eyelid oedema (Eye disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 13
Abdominal pain upper (Gastrointestinal disorders) | 11
Constipation (Gastrointestinal disorders) | 23
Diarrhoea (Gastrointestinal disorders) | 49
Dyspepsia (Gastrointestinal disorders) | 13
Nausea (Gastrointestinal disorders) | 33
Stomatitis (Gastrointestinal disorders) | 12
Vomiting (Gastrointestinal disorders) | 22
Asthenia (General disorders) | 13
Chest pain (General disorders) | 7
Fatigue (General disorders) | 36
Mucosal inflammation (General disorders) | 15
Oedema peripheral (General disorders) | 24
Pain (General disorders) | 8
Pyrexia (General disorders) | 15
Nasopharyngitis (Infections and infestations) | 7
Upper respiratory tract infection (Infections and infestations) | 9
Blood creatinine increased (Investigations) | 8
Weight decreased (Investigations) | 10
Decreased appetite (Metabolism and nutrition disorders) | 27
Hypokalaemia (Metabolism and nutrition disorders) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Back pain (Musculoskeletal and connective tissue disorders) | 18
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11
Dizziness (Nervous system disorders) | 10
Dysgeusia (Nervous system disorders) | 12
Headache (Nervous system disorders) | 20
Cough (Respiratory, thoracic and mediastinal disorders) | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 14
Dry skin (Skin and subcutaneous tissue disorders) | 11
Erythema (Skin and subcutaneous tissue disorders) | 9
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 20
Rash (Skin and subcutaneous tissue disorders) | 9
Hypertension (Vascular disorders) | 16

LIMITATIONS AND CAVEATS:
The reason for not completed 'Study Terminated by Sponsor' in participant flow table indicates the termination of study at few sites as captured in case report forms at those sites and does not reflect overall status of study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.